CLINICAL TRIAL: NCT00250458
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Elimination of Migraine-Associated Nausea in Migraine Patients Treated With Rizatriptan Orally Disintegrating Tablet (ODT)
Brief Title: Study to Test a Marketed Product in the Treatment of Migraine-associated Nausea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0462-074; 2005_081
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Results first posted 2010-06-23 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Rizatriptan (MK0462)10 mg orally disintegrating tablet/oral lyophilisate
  Interventions: Drug: Comparator: Rizatriptan
- 2 (Placebo Comparator): matching placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Comparator: Rizatriptan — One dose Rizatriptan 10 mg orally disintegrating tablet / oral lyophilisate to treat one migraine attack.
  Arms: 1
Drug: Comparator: Placebo — One dose matching placebo to Rizatriptan to treat one migraine attack.
  Arms: 2

SUMMARY:
Study to test the effectiveness of a marketed drug in the treatment of migraine-associated nausea.

ELIGIBILITY:
Inclusion Criteria:

* 6-month history of migraine, moderate to severe migraine attacks with nausea, 1-6 migraine attacks per month

Exclusion Criteria:

* Heart disease, high blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2006-03; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Freitag F, Taylor FR, Hamid MA, Rodgers A, Hustad CM, Ramsey KE, Skobieranda F. Elimination of migraine-associated nausea in patients treated with rizatriptan orally disintegrating tablet (ODT): a randomized, double-blind, placebo-controlled study. Headache. 2008 Mar;48(3):368-77. doi: 10.1111/j.1526-4610.2007.00954.x. Epub 2007 Nov 28. PMID 18047500

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-Four (24) investigators in the United States
  Primary Therapy Period: MAR06 to OCT06.
Pre-assignment Details: Each patient was to treat one migraine attack of moderate or severe intensity with accompanying nausea. Rescue medication was allowed for headache non-response or recurrence after 2 hours postdose. Patients were to treat a qualifying migraine attack within 3 months after randomization.
Groups:
- Rizatriptan 10 mg: Rizatriptan 10 mg Orally Disintegrating Tablet (ODT), one dose, to treat a single migraine attack
- Placebo: Placebo matching Rizatiptan 10 mg ODT, one dose, to treat a single migraine attack
Period: Overall Study
Arm/Group | Rizatriptan 10 mg | Placebo
Started | 232 | 114
Completed | 200 | 97
Not Completed | 32 | 17
Not completed — Lost to Follow-up | 4 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lack of Migraine Attack | 20 | 9
Not completed — Qualifying migraine but did not treat | 3 | 3
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rizatriptan 10 mg | Placebo | Total
Number analyzed (Participants) | 232 | 114 | 346
Age, Continuous [Mean (Full Range); unit: Years] | 40 [18 to 65] | 41 [18 to 60] | 40 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 103 | 310
  Male | 25 | 11 | 36

OUTCOME MEASURES:

1. Primary Outcome: Participants With Elimination of Nausea at 2 Hours Postdose
Description: Participants reporting the absence of nausea at 2 hours post treatment. Absence or presence of nausea was recorded by the participants in an electronic diary. Absence is defined as no nausea at 2 hours post-treatment.
Time Frame: At 2 hours after treatment
Population: Full Analysis Set (FAS): The FAS population included all randomized and treated Participants who had at least one assessment within 2 hours post-dose (i.e., after baseline assessment).
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 10 mg | Placebo
Number analyzed (Participants) | 185 | 92
Participants
  No Nausea at 2 Hours | 130 | 57
  Nausea at 2 Hours | 55 | 35

2. Secondary Outcome: Participants With Pain Relief at 2 Hours Postdose
Description: Participants reporting pain relief defined as a reduction of pain severity from grades 2 or 3 (moderate or severe pain) at baseline to grades 0 or 1 (no headache or mild pain) at 2 hours after treatment.
Time Frame: 2 hours after treatment
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 10 mg | Placebo
Number analyzed (Participants) | 185 | 92
Participants
  2-Hour Pain Relief | 129 | 50
  No 2-Hour Pain Relief | 56 | 42

ADVERSE EVENTS:
Time Frame: Reporting of adverse experiences from the time of informed consent to Visit 2. All serious adverse experiences that occur during this period and up to 14 days postdose of study therapy.
Description: Number of subjects at risk included randomized subjects who had follow-up after at least one dose of study medication.
Arm/Group | Rizatriptan 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/97
Other Adverse Events (participants affected / at risk) | 30/200 | 4/97
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rizatriptan 10 mg (N=200) | Placebo (N=97)
Palpitations (Cardiac disorders) | 1 | 0
Vision blurred (Eye disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Paraesthesia oral (Gastrointestinal disorders) | 2 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 1 | 1
Peripheral coldness (General disorders) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 1
Dysgeusia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 4 | 0
Tremor (Nervous system disorders) | 1 | 0
Dissociative disorder (Psychiatric disorders) | 1 | 0
Euphoric mood (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Pharyngeal hypoaesthesia (Psychiatric disorders) | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.